CLINICAL TRIAL: NCT02415491
Title: Cardiovascular Magnetic Resonance at Rest and Stress in Relation to Cardiopulmonary Exercise Capacity in Young Adults After Arterial Switch Operation (ASO) for Transposition of the Great Arteries (TGA)
Brief Title: Cardiovascular MRI and Cardiopulmonary Exercise Capacity After Neonatal ASO) in Young Adults
Acronym: ASO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-039
Record Dates: First submitted 2015-04-01; First posted 2015-04-14 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Transposition of the Great Arteries; Artery Switch Operation
Keywords: TGA; ASO; magnetic resonance imaging (MRI); young adulthood
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASO group (Experimental): ASO group:Evaluation of Correlation of Heart Magnetic Resonance Imaging at rest and stress with Cardiopulmonary stress test for long term assessment after ASO and recommendation of physical activity of young adults after TGA
  Interventions: Other: Correlation Heart Magnetic Resonance Imaging at rest and stress with Cardiopulmonary stress test

INTERVENTIONS:
Other: Correlation Heart Magnetic Resonance Imaging at rest and stress with Cardiopulmonary stress test — MRI of the heart, coronary arteries and pulmonary artery at rest and stress induced will be performed. Cine pictures are taken for evaluation of pulmonary perfusion.
  Afterwards induced stress MRI will be performed according to standard protocol with elevation of dobutamine levels until the reach of peak HR. If applicable the procedure will be stopped) in case of e.g. arrhythmia.
  Cardiopulmonary exercise stress test will be performed; patient will sit at rest on the ergometer, the subject's gas exchange will be recorded; with the pedal speed constant, the resistance will be increased from 0.5 watt/kg to 3 watt/kg over 10 minutes. Electrocardiography and heart rate will be taken continuously during and until 10 minutes afterwards. Blood pressure will be taken before, during and after the stress test. Respiratory gas exchange parameters will be taken continuously, peak oxygen uptake (VO2) determined as well as Ventilatory Efficiency.

SUMMARY:
Magnetic Resonance Imaging of the heart at rest and stress conditions relative to the cardiopulmonary exercise capacity in young adults after neonatal surgery for transposition of the great arteries.

DETAILED DESCRIPTION:
After ASO obstruction of the transposed coronary arteries with resulting reduced perfusion of the heart at stress or abnormities of the right ventricular blood flow resulting in increasing heart rate as well as abnormities in pulmonary flow can appear. In this single centre trial a large homogeneous group of young adults after surgery for transposition of the great arteries (TGA), the so called artery switch operation (ASO), will undergo magnetic resonance imaging (MRI) of the heart at rest and under drug- induced stress to receive data of the functional status of the heart and its perfusion as well as data of the pulmonary arterial perfusion.

Also obstruction of the pulmonary arteries will lead to reduced perfusion and cardiopulmonary exercise capacity.

Therefore the MRI data will be compared to cardiopulmonary exercise capacity data determined by cardio pulmonary stress test (CPX) concerning the feasibility of a correlation of the data and possible generalisation of the results leading to long term assessment of coronary perfusion and myocardial status after ASO for recommendations of physical activity of the young adults.

ELIGIBILITY:
Inclusion Criteria:

* former EMAH (adults with congenital heart defects) patients > 18 years old
* after neonatal ASO for TGA at the Department of pediatric cardiac surgery
* also if applicable with a correction of an aorta isthmus stenosis neotal or in infancy

Exclusion Criteria:

* contraindications of MRI as metallic implants, claustrophobia
* contraindications of MRI contrast agents
* severe chronic kidney disease (estimated glomerular filtration rate < 30 ml/min)
* contraindications of exercise stress test with dobutamine or cardiopulmonary exercise stress test (e.g. instable angina pectoris, complex arrhythmia)
* disabled persons not able to perform cardiopulmonary exercise stress test
* pregnancy and breast feeding

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction (EF) | up to 3 hours
  MRI of the heart, coronary arteries and pulmonary artery at rest and stress induced will be performed. Cine pictures are taken for evaluation of the ejection fraction.
  Afterwards induced stress MRI will be performed according to standard protocol, with elevation of dobutamine levels every 3 minutes from 10 microgram /kg/min to 40 microgram until the reach of peak HR. If applicable the procedure will be stopped in case of e.g. arrhythmia.
Heart rate (HR) | up to 3 hours
  MRI at rest will be performed, afterwards induced stress MRI will be performed according to standard protocol, with elevation of dobutamine levels every 3 minutes from 10 microgram /kg/min to 40 microgram until the reach of peak HR. If applicable the procedure will be stopped in case of e.g. arrhythmia.
Wall motion | up to 3 hours
  MRI of the heart, coronary arteries and pulmonary artery at rest and stress induced will be performed. Cine pictures are taken for evaluation of wall motions.
  Induced stress MRI will be performed according to standard protocol, with elevation of dobutamine levels every 3 minutes from 10 microgram /kg/min to 40 microgram until the reach of peak HR. If applicable the procedure will be stopped in case of e.g. arrhythmia.
Pulmonary ventilation/pulmonary blood flow (V/Q in l/min) | up to 3 hours
  MRI of the heart, coronary arteries and pulmonary artery at rest and stress induced will be performed. Cine pictures are taken for evaluation of pulmonary perfusion.
  Afterwards induced stress MRI will be performed according to standard protocol with elevation of dobutamine levels every 3 minutes from 10 microgram /kg/min to 40 microgram/kg/min until the reach of peak HR. If applicable the procedure will be stopped in case of e.g. arrhythmia.

SECONDARY OUTCOMES:
Breathing minute volume (VE l/min) | up to 1 hour
  cardiopulmonary exercise stress test will be performed; patient will sit at rest on the ergometer and the subject's gas exchange will be recorded; with the pedal speed constant, the resistance will be increased from 0.5 watt/kg to 3 watt/kg over 10 minutes. Electrocardiography and heart rate will be taken continuously during and until 10 minutes afterwards. Blood pressure will be taken before, during and after the stress test.
Peak oxygen uptake (VO2 in %) | up to 1 hour
  cardiopulmonary exercise stress test will be performed; patient will sit at rest on the ergometer and the subject's gas exchange will be recorded; with the pedal speed constant, the resistance will be increased from 0.5 watt/kg t0 3 watts/kg over 10 minutes. Electrocardiography and heart rate will be taken continuously during and until 10 minutes afterwards. Blood pressure will be taken before, during and after the stress test. Respiratory gas exchange parameters will be taken continuously, peak VO2 determined.
Forced vital capacity (in %) | up to 1 hour
  cardiopulmonary exercise stress test will be performed; patient will sit at rest on the ergometer and the subject's gas exchange will be recorded; with the pedal speed constant, the resistance will be increased from 0.5 watt/kg t0 3 watt/kg over 10 minutes. Electrocardiography and heart rate will be taken continuously during and until 10 minutes afterwards. Blood pressure will be taken before, during and after the stress test. Respiratory gas exchange parameters will be taken, forced vital capacity determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hedwig Hoevels-Guerich, Prof MD, Principal Investigator — Department od Pediatric Cardiology, University Hospital Aachen
Locations (1):
- University Hospital Aachen, Department od Pediatric Cardiology, Aachen, Germany